CLINICAL TRIAL: NCT04302870
Title: Motor Neurone Disease - Systematic Multi-Arm Adaptive Randomised Trial
Acronym: MND-SMART
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: University College, London (Other); University of Warwick (Other); NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC18082
Record Dates: First submitted 2020-03-04; First posted 2020-03-10 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2024-12

CONDITIONS: Motor Neuron Disease, Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Memantine; Trazodone; Amantadine; Tacrolimus; Capsules

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Memantine (Experimental)
  Interventions: Drug: Memantine Hydrochloride Oral Solution
- Trazodone (Experimental)
  Interventions: Drug: Trazodone Hydrochloride oral solution
- Placebo (liquid) (Placebo Comparator)
  Interventions: Drug: Placebo oral solution
- Amantadine (Experimental)
  Interventions: Drug: Amantadine Hydrochloride Oral Solution
- Tacrolimus (Experimental)
  Interventions: Drug: Tacrolimus 1Mg Cap
- Placebo (tablet) (Placebo Comparator)
  Interventions: Drug: Placebo capsule

INTERVENTIONS:
Drug: Memantine Hydrochloride Oral Solution — Memantine hydrocholoride taken once daily
  Arms: Memantine
Drug: Trazodone Hydrochloride oral solution — Trazodone Hydrochloride taken once daily
  Arms: Trazodone
Drug: Placebo oral solution — Placebo taken once daily
  Arms: Placebo (liquid)
Drug: Amantadine Hydrochloride Oral Solution — Amantadine Hydrochloride taken once daily
  Arms: Amantadine
Drug: Tacrolimus 1Mg Cap — Tacrolimus 1Mg overencapsulated tablet taken once daily
  Arms: Tacrolimus
Drug: Placebo capsule — Placebo taken once daily
  Arms: Placebo (tablet)

SUMMARY:
MND-SMART is investigating whether selected drugs can slow down the progression of motor neuron disease (MND) and improve survival.

The study is 'multi-arm' meaning more than one treatment will be tested at the same time. The trial started with 3 arms; drug 1 (memantine), drug 2 (trazodone) and placebo (dummy drug). A third drug, amantadine, was added in April 2023. A fourth drug, tacrolimus, was added in March 2025 in Edinburgh and across all sites in April 2025. The first two drugs, memantine and trazodone, were removed from the trial in September 2023 due to lack of benefit. The trial currently has 4 recruiting arms; amantadine, liquid placebo (matched to amantadine), tacrolimus, and tablet placebo (matched to tacrolimus). This allows the evaluation of each drug versus placebo. Participants will be randomly allocated between the treatment arms they are eligible for. Medicines being tested are already approved for use in other conditions.

MND-SMART has an 'adaptive' design. This means medicines being studied can change according to emerging results. Treatments shown to be ineffective can be dropped and new drugs can be added over the duration of the study. This will allow many treatments, over time, to be efficiently and definitively evaluated.

The medicines being tested have been selected following a rigorous process involving a systematic, unbiased, and comprehensive review of past clinical trials data, as well as information from pre-clinical research (studies in laboratories), for MND and other related neurodegenerative disorders. Drugs have been ranked for inclusion in MND-SMART by a group of independent MND experts according to set criteria. These include consideration of how the drugs work, their safety profiles, and the quality of previous studies.

New drugs will be selected for investigation in MND-SMART based on continuous review of constantly updated scientific evidence as well as findings from state-of-the-art human stem cell based drug discovery platforms. These can be added by substantial amendment to the protocol.

DETAILED DESCRIPTION:
For further information, please visit: https://mnd-smart.org/

ELIGIBILITY:
Participants will be considered eligible for randomisation if they fulfil all the core inclusion criteria and none of the exclusion criteria as defined below. In addition, investigators must simultaneously check and ensure participants do not meet any of the drug specific exclusion criteria. If exclusion criteria are met for an arm, participants can still be considered for other arms and randomised accordingly to eligible arms.

Core inclusion criteria:

* Confirmed diagnosis of MND. This includes the following subtypes: ALS by El Escorial Criteria (possible, probable, and definite) or Gold Coast Criteria, Primary Lateral Sclerosis, and Progressive Muscular Atrophy
* Over 18
* Women of childbearing potential according to CTFG guidelines must have a negative pregnancy test within 7 days prior to, or at, the baseline visit
* Women of childbearing potential and fertile men must be using an appropriate method of contraception to avoid any unlikely teratogenic effects of the selected drugs from time of consent, to 4 weeks after treatment inclusive
* Willing and able to comply with the trial protocol and ability to understand and complete questionnaires
* Written informed consent (in the case of limb dysfunction verbal consent can be given in the presence of a witness who can sign)

Core Exclusion Criteria:

* Patients diagnosed with Frontotemporal Dementia (FTD-MND) or any other significant psychiatric disorder that prevents informed consent being given.
* Alcoholism (current self-reported - at the investigator's discretion)
* Active suicide ideation assessed using the Columbia-Suicide Severity Rating Scale
* On concurrent investigational devices and medication (including biological therapy)
* Pregnancy or breast-feeding females
* If ALT, ALP, bilirubin or GGT >3 times the upper limit of normal.
* If creatinine clearance (creatinine clearance or eGFR) <35 ml/min.
* If TSH <0.2mU/l (if possible to test free T4, then Serum free T4 >25pmol/l)
* If corrected QT interval on 12 lead ECG >500 ms
* Patient's diagnosed with ventricular arrhythmias, significant heart block (at the investigator's discretion)) or in the immediate recovery period after myocardial infarction (< 6 weeks).
* Patients who the PI considers will not be able to comply with the study protocol.

Amantadine Exclusion Criteria:

* Patients in the manic phase of bipolar disorder.
* Patients with history of proven peptic ulcer confirmed on endoscopy
* Patients with active epilepsy
* Already taking the IMP in this comparison
* Known hypersensitivity, including hereditary fructose intolerance, or adverse reaction to the active substances and their excipients (as per SPCs for this comparison) or any past medical history contraindicating use of the IMP in this comparison

Tacrolimus Exclusion Criteria:

* Poorly controlled hypertension (Systolic BP>180 mmHg or Diastolic BP>100mmHg)
* Poorly controlled diabetes (HbA1c>6.4% or 48mmol/mol)
* Hypertrophic cardiomyopathy or history of QT prolongation (including family history), congestive heart failure, bradyarrhythmias, and electrolyte abnormalities
* History of bleeding disorders or significant haematological or immune diseases including, congenital or acquired immune deficiency, anaemia (Hb<130g/L for males and Hb<120 g/L in females) and thrombocytopenia (platelet count <150 × 109/L), use of other biological agents and immunosuppressant medications including oral/IV steroids
* Active or chronic infection (at PI discretion)
* History of Hepatitis B or C
* History of lymphoma and active malignancy
* Risk of dehydration due to reduced oral intake and lack of parenteral route
* Patient's contraindicated to tacrolimus according to SPC section 4.3
* Use of concomitant medications that interacts with tacrolimus according to the SPC, including but not limited to strong CYP3A4 inhibitors (i.e. azoles, protease inhibitors) or CYP3A4 inducers (rifampicin, phenytoin, carbamazepine), barbiturates, macrolides, digoxin, statins, PPI inhibitors, ergotamine, tricyclic antidepressants, herbal supplements (St. John's wort, extracts of Schisandra sphenanthera)
* Inability to swallow capsules
* Already taking the IMP in this comparison
* Known hypersensitivity, including lactose and gelatin intolerance, or adverse reaction to the active substances and their excipients (as per SPCs for this comparison) or any past medical history contraindicating use of the IMP in this comparison
* Receipt of a live attenuated vaccine within four weeks prior to receipt of tacrolimus. These include, but are not limited to live influenza vaccine (Fluenz Tetra), Shingles (varicella zoster virus) Zostavax, Varicella (Varilrix, Varilvax), Oral typhoid (Ty21a), and yellow fever vaccines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1150 (Estimated)
Dates: Start 2020-02-27 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Change in decline of ALS-FRS(R) over 18months | 18 months
  Co-primary outcome measure
Survival | 18 months
  Co-primary outcome measure

SECONDARY OUTCOMES:
Cognition and behaviour | 18 months
  Using Edinburgh Cognitive and Behavioural ALS Screen (ECAS)
Respiratory function - Forced vital capacity | 18 months
  Change in FVC
King's ALS Clinical stage | 18 months
  Time to reach King's stage IV, scale range I - V
Changes in anxiety and depression | 18 months
  Measured using the hospital anxiety and depression scale (HADS), scale range 0 - 42
Changes in Quality of Life | 18 months
  Measured using EQ-5D-5L
Safety and tolerability of IMPs | 18 months
  Measured using adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Professor Chandran, Study Director — University of Edinburgh
Locations (22):
- United Kingdom (22):
  - Southern Health and Social Care Trust, Craigavon Area Hospital, Portadown, County Armagh
  - Aberdeen Royal Infirmary, Aberdeen
  - University Hospitals of Birmingham NHS Foundation Trust, Birmingham
  - University Hospitals Sussex NHS Foundation Trust, Brighton
  - West Suffolk NHS Foundation Trust, Bury St Edmunds
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Cardiff and Vale University Local Health Board, Cardiff
  - Clinical Research Centre , Ninewells Hospital, Dundee
  - Anne Rowling Regenerative Neurology Clinic, Edinburgh
  - Royal Devon and Exeter Hospital, Exeter
  - Queen Elizabeth University Hospital Clinical Research Facility, Glasgow
  - NHS Highland Clinical Research Facility, Raigmore Hospital, Inverness
  - East Suffolk and North Essex NHS Foundation Trust, Ipswich
  - Royal London Hospital, London
  - St George's University Hospitals NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich
  - University Hospitals of Dorset NHS Trust, Poole
  - Clinical Research Facility Salford Royal NHS Foundation Trust, Salford
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - Clinical Research Facility University Hospital Southampton, Southampton

IPD SHARING:
Plan to Share IPD: Yes
To ensure data transparency, the results of any closed comparisons will be published in a peer reviewed journal as soon as it is possible when the integrity of the trial will not be affected.
  Individual level participant data will be shared ,after deidentification, upon receipt of a valid request.
  Some data may be shared prior to the publication of study results depending on the requirements, however no end point data will be released without explicit need and permission from the TSC.
  Each data request form will be individually reviewed to ensure the proposal has a valid rationale and appropriate methodology. Only data required for the project will be shared.
  A summary of results will be provided to all participants via newsletters and the trial website.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After publication of study results, no end date.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal to achieve the aims of the proposal only.
  Data sharing request forms are available from mnd-smart@Ed.ac.uk. Requesters will need to sign a data access agreement prior to being provided with access to data.

REFERENCES:
- [Derived] Pal S, Chataway J, Swingler R, Macleod MR, Carragher NO, Hardingham G, Selvaraj BT, Smith C, Wong C, Newton J, Lyle D, Stenson A, Dakin RS, Ihenacho A, Colville S, Mehta AR, Stallard N, Carpenter JR, Parker RA, Keerie C, Weir CJ, Virgo B, Morris S, Waters N, Gray B, MacDonald D, MacDonald E, Parmar MKB, Chandran S; MND SMART Investigators. Safety and efficacy of memantine and trazodone versus placebo for motor neuron disease (MND SMART): stage two interim analysis from the first cycle of a phase 3, multiarm, multistage, randomised, adaptive platform trial. Lancet Neurol. 2024 Nov;23(11):1097-1107. doi: 10.1016/S1474-4422(24)00326-0. Epub 2024 Sep 19. PMID 39307154
- [Derived] Wong C, Gregory JM, Liao J, Egan K, Vesterinen HM, Ahmad Khan A, Anwar M, Beagan C, Brown FS, Cafferkey J, Cardinali A, Chiam JY, Chiang C, Collins V, Dormido J, Elliott E, Foley P, Foo YC, Fulton-Humble L, Gane AB, Glasmacher SA, Heffernan A, Jayaprakash K, Jayasuriya N, Kaddouri A, Kiernan J, Langlands G, Leighton D, Liu J, Lyon J, Mehta AR, Meng A, Nguyen V, Park NH, Quigley S, Rashid Y, Salzinger A, Shiell B, Singh A, Soane T, Thompson A, Tomala O, Waldron FM, Selvaraj BT, Chataway J, Swingler R, Connick P, Pal S, Chandran S, Macleod M. Systematic, comprehensive, evidence-based approach to identify neuroprotective interventions for motor neuron disease: using systematic reviews to inform expert consensus. BMJ Open. 2023 Feb 1;13(2):e064169. doi: 10.1136/bmjopen-2022-064169. PMID 36725099
- [Derived] Parker RA, Weir CJ, Pham TM, White IR, Stallard N, Parmar MKB, Swingler RJ, Dakin RS, Pal S, Chandran S. Statistical analysis plan for the motor neuron disease systematic multi-arm adaptive randomised trial (MND-SMART). Trials. 2023 Jan 16;24(1):29. doi: 10.1186/s13063-022-07007-z. PMID 36647114
- [Derived] Wong C, Dakin RS, Williamson J, Newton J, Steven M, Colville S, Stavrou M, Gregory JM, Elliott E, Mehta AR, Chataway J, Swingler RJ, Parker RA, Weir CJ, Stallard N, Parmar MKB, Macleod MR, Pal S, Chandran S. Motor Neuron Disease Systematic Multi-Arm Adaptive Randomised Trial (MND-SMART): a multi-arm, multi-stage, adaptive, platform, phase III randomised, double-blind, placebo-controlled trial of repurposed drugs in motor neuron disease. BMJ Open. 2022 Jul 7;12(7):e064173. doi: 10.1136/bmjopen-2022-064173. PMID 35798516